CLINICAL TRIAL: NCT05145192
Title: Validity and Reliability of the K5 Wearable Metabolic System During High-Intensity Treadmill Testing in Healthy, Young Adults
Brief Title: COSMED K5 Validation and Reliability Study
Acronym: K5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Simon Driver, Research Center Director - The STAR at Frisco, Baylor Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 021-348
Record Dates: First submitted 2021-11-17; First posted 2021-12-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Cardiopulmonary; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- COSMED K5 CPET (Experimental): Participants in this arm will complete the CPET using the COSMED K5 wearable metabolic system at first visit and the ParvoMedics TrueOne® 2400 automated metabolic gas analysis system at second visit.
  Interventions: Device: COSMED K5 CPET (Cardiopulmonary Exercise Test); Device: ParvoMedics CPET
- ParvoMedics CPET (Active Comparator): Participants in this arm will complete the CPET using the ParvoMedics TrueOne® 2400 automated metabolic gas analysis system at first visit and the COSMED K5 wearable metabolic system at second visit.
  Interventions: Device: COSMED K5 CPET (Cardiopulmonary Exercise Test); Device: ParvoMedics CPET

INTERVENTIONS:
Device: COSMED K5 CPET (Cardiopulmonary Exercise Test) — In this randomized crossover trial of eligible adults, we will compare peak measurements of oxygen consumption (VO2) and carbon dioxide production (VCO2) during three maximal cardiopulmonary stress exercise tests (CPET), each seven to ten days apart. Subjects will be randomized into either the K5 or ParvoMedics (PM) group for their first CPET using a 1:1 randomization scheme and will serve as their own control in the subsequent test seven to ten days after the previous one. After both a K5 and a PM CPETs have been completed, the participants will complete an additional K5 CPET for test-retest reliability. A within-subjects analysis will be performed.
Device: ParvoMedics CPET — ParvoMedics CPET

SUMMARY:
To determine the validity of the K5 metabolic system breath-by-breath analysis setting during a high intensity treadmill running protocol compared to the criterion ParvoMedics TrueOne® 2400 automated metabolic gas analysis system.

To determine the test-retest reliability of the K5 metabolic system breath-by-breath analyzer during a high intensity treadmill protocol (Bruce Protocol).

ELIGIBILITY:
Inclusion Criteria:

* 20-29 years of age

Exclusion Criteria:

* Pregnancy
* Children
* Inmates
* Neuromotor, musculoskeletal, or rheumatoid disorders that are exacerbated by exercise or conditions preventing cooperation
* Contraindications to Symptom-limited Maximal Exercise Testing
* Metabolic disease
* Pacemakers/Implantable devices
* Supplemental Oxygen use
* Diagnosis of severe arterial hypertension
* Uncontrolled asthma

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption (VO2), mL/min | At first assessment, during week one.
  Using metabolic cart, VO2 will be recorded.
Oxygen consumption (VO2), mL/min | At second assessment, during week two.
  Using metabolic cart, VO2 will be recorded.
Oxygen consumption (VO2), mL/min | At third assessment, during week three.
  Using metabolic cart, VO2 will be recorded.
Carbon dioxide production (VCO2), mL/min | At first assessment, during week one.
  Using metabolic cart, VCO2 will be recorded.
Carbon dioxide production (VCO2), mL/min | At second assessment, during week two.
  Using metabolic cart, VCO2 will be recorded.
Carbon dioxide production (VCO2), mL/min | At third assessment, during week three.
  Using metabolic cart, VCO2 will be recorded.

SECONDARY OUTCOMES:
Respiratory Exchange Ratio (RER) | At first assessment, during week one.
  Using metabolic cart, respiratory exchange ratio will be recorded.
Respiratory Exchange Ratio (RER) | At second assessment, during week two.
  Using metabolic cart, respiratory exchange ratio will be recorded.
Respiratory Exchange Ratio (RER) | At third assessment, during week three.
  Using metabolic cart, respiratory exchange ratio will be recorded.
Minute Ventilation, L/min | At first assessment, during week one.
  Using metabolic cart, minute ventilation will be recorded.
Minute Ventilation, L/min | At second assessment, during week two.
  Using metabolic cart, minute ventilation will be recorded.
Minute Ventilation, L/min | At third assessment, during week three.
  Using metabolic cart, minute ventilation will be recorded.
Breathing Reserve, % | At first assessment, during week one.
  Using metabolic cart, breathing reserve will be recorded.
Breathing Reserve, % | At second assessment, during week two.
  Using metabolic cart, breathing reserve will be recorded.
Breathing Reserve, % | At third assessment, during week three.
  Using metabolic cart, breathing reserve will be recorded.
Tidal Volume, L | At first assessment, during week one.
  Using metabolic cart, tidal volume will be recorded.
Tidal Volume, L | At second assessment, during week two.
  Using metabolic cart, tidal volume will be recorded.
Tidal Volume, L | At third assessment, during week three.
  Using metabolic cart, tidal volume will be recorded.
Respiratory Frequency, /min | At first assessment, during week one.
  Using metabolic cart, respiratory frequency will be recorded.
Respiratory Frequency, /min | At second assessment, during week two.
  Using metabolic cart, respiratory frequency will be recorded.
Respiratory Frequency, /min | At third assessment, during week three.
  Using metabolic cart, respiratory frequency will be recorded.
Fractional expired oxygen (FEO2) | At first assessment, during week one.
  Using metabolic cart, fractional expired oxygen will be recorded.
Fractional expired oxygen (FEO2) | At second assessment, during week two.
  Using metabolic cart, fractional expired oxygen will be recorded.
Fractional expired oxygen (FEO2) | At third assessment, during week three.
  Using metabolic cart, fractional expired oxygen will be recorded.
Fractional expired carbon dioxide (FECO2) | At first assessment, during week one.
  Using metabolic cart, fractional expired carbon dioxide will be recorded.
Fractional expired carbon dioxide (FECO2) | At second assessment during week two.
  Using metabolic cart, fractional expired carbon dioxide will be recorded.
Fractional expired carbon dioxide (FECO2) | At third assessment, during week three .
  Using metabolic cart, fractional expired carbon dioxide will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott and White Sports Therapy and Research, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No